CLINICAL TRIAL: NCT04389216
Title: Radiofrequency Ablation in Breast Tumors in Early Stages
Brief Title: Radiofrequency Ablation (RFA) in Breast Tumors
Acronym: RFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Amparo Garcia-Tejedor, PRINCIPAL INVESTIGATOR, Hospital Universitari de Bellvitge
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICPS002/20
Record Dates: First submitted 2020-05-03; First posted 2020-05-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Female
Keywords: radiofrequency; early stage
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Radiofrequency ablation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Radiofrequency Ablation Tumor (Experimental): Radiofrequency Ablation of breast cancer tumour by Cool-tip electrode.
  Interventions: Device: Cool-tip electrode for Radiofrequency Ablation

INTERVENTIONS:
Device: Cool-tip electrode for Radiofrequency Ablation — Radiofrequency ablation of the tumour in the surgery group, associated whith axillary surgery when applicable

SUMMARY:
To validate the efficacy and safety of the cool-tip ablation method for breast tumors smaller than 2 cm.

DETAILED DESCRIPTION:
A prospective, phase II-III study, which will include a series of cases of 30 patients. The hospitals involved will be Bellvitge University Hospital and Hospital del Mar.

Efficacy was evaluated according magnetic resonance image and biopsy of the breast 1 month after the procedure.

Patients will be followed up over a 2-year period to assess cosmetic results, short and long-term complications and possible recurrences.

ELIGIBILITY:
Inclusion Criteria:

* Infiltrating ductal carcinoma according the biopsy of the breast,
* Tumor visible by ultrasound, smaller than 2 cm,
* Located > 1 cm from the chest wall and the skin.

Exclusion Criteria:

* Personal antecedents of breast cancer
* Multifocality or intraductal carcinoma
* Lobular infiltrating carcinoma
* Neoadjuvant therapy

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
MRI post-RFA | "1 month"
  Magnetic Resonance Image after Radiofrequency ablation to confirmate complete disappearance of tumor contrast enhancement (residual mm).
BAG post-RFA | "1 month"
  Breast biopsy after Radiofrequency to confirmate absence of viable tumor tissue using NADH, CK18 and CK19 stainings (tumor viability scale: 0, <25%, 25-50%, 50-75%, > 75%).

SECONDARY OUTCOMES:
Adverse Effects | "1 month"
  Adverse effects related to radiofrequency
Quality | "1 month"
  Breast-Q

CONTACTS AND LOCATIONS:
Overall Officials: Amparo Garcia-Tejedor, MDPhD, Principal Investigator — Hospital Universitari Bellvitge
Locations (2):
- Spain (2):
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona

IPD SHARING:
Plan to Share IPD: No